CLINICAL TRIAL: NCT05147506
Title: A Single-Blind, Randomized, Controlled Trial of a Cognitive-Behavioral Therapy Digital Therapeutic to Combat Symptoms of Depression in Service Members and Adults With a History of MildTraumatic Brain Injury
Brief Title: Digital Therapeutic for Depression After Head Injury in Current and Former US Military Personnel
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNRM-92-10531
Record Dates: First submitted 2021-07-20; First posted 2021-12-07 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Depressive Symptoms; Mild Traumatic Brain Injury
MeSH Terms: conditions — Depression; Brain Concussion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CBT DTx (Experimental): Participants randomized to active intervention will access a structured, cognitive behavioral therapy (CBT) intervention.
  Interventions: Device: CNRM DTx
- Psychoeducations DTx (Active Comparator): Participants randomized to the comparison group will access an unstructured educational DTx.
  Interventions: Other: Psychoeducation Comparison

INTERVENTIONS:
Device: CNRM DTx — A mobile application intervention adapted from the CBT for Depression and CBT for TBI manuals.
  Arms: CBT DTx
Other: Psychoeducation Comparison — A mobile application that consists of psychoeducational material regarding depression and brain injury.
  Arms: Psychoeducations DTx

SUMMARY:
The Center for Neuroscience and Regenerative Medicine (CNRM) Clinical Trials Unit has developed the first cognitive-behavioral therapy (CBT) digital therapeutic (DTx) mobile application to counteract depressive symptoms in military service members and veterans with a history of mild traumatic brain injury (mTBI). This trial will assess the efficacy of the novel CBT-DTx for depression following mTBI compared to an educational comparison DTx.

DETAILED DESCRIPTION:
This trial is a single-blind, randomized, controlled interventional trial of current and former military personnel with symptoms of depression and a history of mTBI. The study will be conducted remotely.

ELIGIBILITY:
Inclusion Criteria:

* Be aged ≥ 18 to ≤ 65 years
* Be able to provide informed consent
* Diagnosed with mild TBI as defined by the Department of Veteran's Affairs and Department of Defense Clinical Practice
* Have a PHQ-9 score of ≥ 5 to 27, indicative of mild or greater depressive symptoms
* Have ownership of or reliable access to a smartphone with a data plan or internet connecting capabilities
* While participating in this study, be able to ensure that you have access to regular care for mental health and to speak with your provider as necessary

Exclusion Criteria:

* Report of starting pharmacological or non-pharmacological treatment for depression within the 3 months prior to trial enrollment
* Report a recent change in type or dose of antidepressant medications within 12 weeks prior to trial enrollment
* Report active psychotic or bipolar symptoms
* Active plan and/or intent of suicide or homicide
* In the opinion of the investigator, they have other considerations that may adversely affect patient safety, participation, or scientific validity of the data being collected

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change of the mean difference in Patient Health Questionnaire (PHQ-9) total score | Week 12 and Week 16 compared to Baseline
  Self-report measure of depression symptom severity; range 0-27; higher score indicates greater severity
Change of the mean difference in Patient Health Questionnaire (PHQ-9) total scores of participants who complete all treatment modules compared to those who do not | Week 12 compared to Baseline
  Self-report measure of depression symptom severity; range 0-27; higher score indicates greater severity
Change of the mean difference in Patient Health Questionnaire (PHQ-9) total scores of participants who report history of depression prior to mTBI compared to those who do not | Week 12 compared to Baseline
  Self-report measure of depression symptom severity; range 0-27; higher score indicates greater severity
Change of the mean difference in Patient Health Questionnaire (PHQ-9) total scores of participants who report family history of depression compared to those who do no | Week 12 compared to Baseline
  Self-report measure of depression symptom severity; range 0-27; higher score indicates greater severity
Change of the mean difference in Patient Health Questionnaire (PHQ-9) total scores, comparison between depression severity group | Week 12 compared to Baseline
  Self-report measure of depression symptom severity; range 0-27; higher score indicates greater severity

SECONDARY OUTCOMES:
Change of the mean difference in Traumatic Brain Injury-Quality of Life (TBI-QOL) total score | Week 12 and Week 16, compared to Baseline
  Computerized adaptive test that measures post-concussive symptoms and quality of life across multiple domains
Change of the mean difference in Posttraumatic Stress Disorder Checklist (PCL-5) total score | Week 12 and Week 16, compared to Baseline
  Self-report measure of PTSD severity; range 0-80; higher score indicates greater severity
Change of the mean difference in Insomnia Severity Index (ISI) total score | Week 12 and Week 16, compared to Baseline
  Self-report measure of insomnia severity; range 0-28; higher score indicates greater severity
Change in Credibility and Expectancy Questionnaire (CEQ) | Week 12 and Week 16, compared to Baseline
  Self-report measure of participation expectation of benefit
Blinding Efficacy | Week 12 and Week 16, compared to Baseline
  Participant blinding questionnaire

OTHER OUTCOMES:
User Version of the Mobile Application Rating Scale (uMARS) | Week 12
  Self-report measure that assess user opinion in 4 objective quality subscales: engagement, functionality, aesthetics, information quality; 1 subjective quality subscale; and 1 scale that measures the perceived impact of the app being evaluated
Mobile Agnew Relationship Measure (mARM) Questionnaire | Week 12
  Self-report measure of therapeutic alliance with mobile health intervention
HEXACO Personality Inventory-Revised (HEXACO-PI-R) | Baseline
  Self-report personality inventory that measures 6 dimensions of personality: honesty-humility, emotionality, eXtraversion, agreeableness (versus anger), conscientiousness, openness to experience

CONTACTS AND LOCATIONS:
Overall Officials: David Brody, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Remote Recruitment: Center for Neuroscience and Regenerative Medicine, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifier-free participant data sets will be shared with the Uniformed Services University Center for Neuroscience and Regenerative Medicine Data Repository. Identifier-free data sets may also be shared with the Federal Interagency Traumatic Brain Injury Research (FITBIR) Data Repository.
Time Frame: After study completion, data sets will be de-identified and shared with the repositories. De-identified data sets will be stored in the repositories indefinitely.
Access Criteria: Access to the CNRM Data Repository will be determined b the CNRM Data Quality, Access, and Publication Committee. Investigators requesting access to the data will provide a list of investigators and collaborators who will have access to the data, documentation of Ethical Conduct of Research and Human Participants Protection Training, and documentation of Institutional Review Board Approval of the research project.
  Access to FITBIR will follow FITBIR Access Criteria
URL: http://fitbir.nih.gov/content/access-data